CLINICAL TRIAL: NCT06596187
Title: Differential Assessment of Hypertonia Related to CNS Impairment
Brief Title: Differential Assessment of Hypertonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SCI_PD_001
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: SCI - Spinal Cord Injury; PD - Parkinson's Disease
Keywords: Spasticity; Post activation depression; Passive motion device (CPM); Rigidity
MeSH Terms: conditions — Spinal Cord Injuries; Parkinson Disease; Muscle Spasticity; Muscle Rigidity | interventions — carboxypeptidase M

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Participants (Experimental): To establish the relationship between changes in foot pressure during ankle joint movement, muscle tone, and Post-Activation Depression (PAD).
  Interventions: Procedure: Continuous passive motion device (CPM) of ankle - fast; Procedure: Continuous passive motion device (CPM) of ankle - slow
- PD Patients (Experimental): To establish the relationship between changes in foot pressure during ankle joint movement, muscle tone, and Post-Activation Depression (PAD).
  Interventions: Procedure: Continuous passive motion device (CPM) of ankle - fast; Procedure: Continuous passive motion device (CPM) of ankle - slow
- SCI Patients (Experimental): To establish the relationship between changes in foot pressure during ankle joint movement, muscle tone, and Post-Activation Depression (PAD).
  Interventions: Procedure: Continuous passive motion device (CPM) of ankle - fast; Procedure: Continuous passive motion device (CPM) of ankle - slow

INTERVENTIONS:
Procedure: Continuous passive motion device (CPM) of ankle - fast — Continuous passive motion device (CPM) of ankle at 1HZ(60rpm) for 10 repetitions
  Other Names: fast CPM
Procedure: Continuous passive motion device (CPM) of ankle - slow — Continuous passive motion device (CPM) of ankle 0.25HZ (15rpm) for 10 repetitions
  Other Names: slow CPM

SUMMARY:
Spasticity and rigidity are common symptoms of central nervous system injuries, such as spinal cord injury and Parkinson's disease, and result in distinct patterns of increased resistance during passive joint movements. Spasticity is characterized by a velocity-dependent increase in stretch reflexes, accompanied by exaggerated tendon responses, while rigidity is marked by consistent resistance throughout the range of motion, traditionally considered independent of stretch velocity. However, recent studies suggest that rigidity may also be influenced by stretch velocity. This study aims to investigate muscle tone by examining spasticity, rigidity, and normal muscle function through neural and biomechanical changes. Standard clinical tools, such as the Modified Ashworth Scale and Unified Parkinson's Disease Rating Scale, along with additional assessments like the Myoton and Post-Activation Depression (PAD), will be employed.

DETAILED DESCRIPTION:
Spasticity and rigidity are common symptoms resulting from central nervous system injuries (e.g., spinal cord injury and Parkinson's disease). During passive joint movement, spasticity and rigidity manifest as two distinct patterns of increased resistance. Spasticity is a type of hypertonia characterized by a stretch reflex that increases with speed, accompanied by exaggerated tendon reflexes. Rigidity, on the other hand, is another form of hypertonia, where resistance increases during passive movement and remains consistent throughout the range of motion.

The degree of rigidity is traditionally considered independent of stretch velocity, which is one of the key differences from spasticity. However, recent studies have found that rigidity may also increase with stretch velocity. Despite attempts to distinguish different types of hypertonia based on stretch velocity, these efforts have largely been unsuccessful. Many factors influence muscle tone, which can be broadly categorized into changes in neural and biomechanical properties. The Modified Ashworth Scale and the Unified Parkinson's Disease Rating Scale are the most commonly used clinical tools for assessing spasticity and rigidity. Additionally, devices such as the Myoton or laboratory parameters like Post-Activation Depression (PAD) are also used for assessment.

ELIGIBILITY:
Health subjects:

Exclusion Criteria:

1. Musculoskeletal injuries on legs.
2. Osteoporosis.

SCI subjects:

Inclusion Criteria 1. Participants with chronic spinal cord injury, with injury duration greater than one year.

Exclusion Criteria

1. Current musculoskeletal or joint injuries in the lower limbs.
2. History of central or peripheral neuromuscular diseases.
3. Presence of a pacemaker.
4. Current use of antispastic or antidepressant medications.
5. Current venous thromboembolism or osteoporosis.
6. Impairment of the soleus H-reflex arc.

PD subjects:

Inclusion Criteria:

- Clinical diagnosis of Parkinson disease.

Exclusion Criteria:

1. Musculoskeletal injuries on legs
2. Osteoporosis.
3. Any peripheral or central nervous system injury or disease patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
H-reflex Amplitude | Before CPM, immediately after CPM
  The peak-to-peak amplitude of the H-reflex measured in the soleus muscle to assess spinal motor neuron excitability. Unit: Millivolts (mV)
M-wave Amplitude | Before CPM, immediately after CPM
  The peak-to-peak amplitude of the M-wave recorded in the soleus muscle to assess peripheral motor neuron excitability and muscle response. Unit: Millivolts (mV)
Level of Post-Activation Depression (PAD) of the H-reflex. | Before CPM, immediately after CPM
  The H-reflex will be elicited by electrical stimulation of the tibial nerve (or other motor nerves), and PAD will be assessed by measuring the reduction in H-reflex amplitude following a series of repetitive stimuli. The amplitude of the H-reflex after repeated stimulation will be compared to the baseline single stimulus.
H/M ratio | Before CPM, immediately after CPM
  The H/M ratio is calculated by dividing the amplitude of the H-reflex by the amplitude of the M-wave.
Muscle Tone (Frequency, Hz) | Before CPM, immediately after CPM
  This parameter measures the natural oscillation frequency of the muscle in response. It reflects the muscle's state of tension or readiness
Elasticity (Dynamic Stiffness, N/m) | Before CPM, immediately after CPM
  Elasticity, measured in Newtons per meter, reflects the muscle's ability to return to its original shape after being deformed by the impulse
Stiffness (Decay, ms) | Before CPM, immediately after CPM
  This parameter quantifies the rate at which the muscle returns to its initial state after the impulse, indicating the muscle's stiffness.
Mechanical Stress (Creep, s) and Relaxation (S) | Before CPM, immediately after CPM
  These parameters measure the time it takes for muscle tissue to adapt to a sustained force (creep) and the time it takes for the muscle to return to a relaxed state after removing the force (relaxation)
Plantar foot pressure distribution and peak pressure | Measured continuously during CPM
  Foot pressure will be measured using a pressure sensors during ankle movement.

SECONDARY OUTCOMES:
M-wave Latency | Before CPM, immediately after CPM
  The time from the onset of electrical stimulation to the onset of the M-wave response in the soleus muscle, used to assess changes in peripheral nerve conduction velocity. Unit: Milliseconds (ms)

OTHER OUTCOMES:
Muscle spasticity levels as assessed by the Modified Ashworth Scale (MAS). | Baseline
  Muscle spasticity levels will be assessed using the Modified Ashworth Scale (MAS), which evaluates resistance during passive soft-tissue stretching. This measure will be used to evaluate changes in muscle tone before and immediately after the intervention. Unit: MAS score (ordinal scale from 0 to 4, where 0 indicates no increase in muscle tone and 4 indicates rigidity in flexion or extension)
Overall the Parkinson's Disease Questionnaire-39 (PDQ-39) Score | Baseline
  An aggregated score derived from the eight dimension scores, providing a comprehensive measure of the individual's quality of life.
Overall the Patient Reported Impact of Spasticity Measure(PRISM) Score | Baseline
  : An aggregated score derived from all the individual items within the questionnaire, providing a comprehensive measure of the impact of spasticity on the patient's quality of life.
Total The Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score | Baseline
  The sum of scores from all 14 items, providing an overall measure of motor impairment severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan